CLINICAL TRIAL: NCT05799157
Title: Protocol 250-1951-201: A Phase 2, Multi-Center, Randomized, Double-Blind, Vehicle-Controlled Study of the Safety and Efficacy of VDMN-21 in Subjects With Verruca Vulgaris
Brief Title: Safety and Efficacy of VDMN-21 Patch in Subjects With Common Warts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Veradermics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 250-12951-201
Record Dates: First submitted 2023-03-22; First posted 2023-04-05 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Verruca Vulgaris; Warts; Common Wart
MeSH Terms: conditions — Warts

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment Group A (Low Dose) (Experimental): Low does patch will be applied adjacent to the target wart and remain in place for 5 minutes then removed. There may be up to 6 treatments (approximately 1 per month).
  Interventions: Drug: VDMN-21 Patch Low Dose
- Treatment Group B (High Dose) (Experimental): High does patch will be applied adjacent to the target wart and remain in place for 5 minutes then removed. There may be up to 6 treatments (approximately 1 per month).
  Interventions: Drug: VDMN-21 Patch High Dose
- Treatment Group C (Vehicle) (Placebo Comparator): Vehicle patch will be applied adjacent to the target wart and remain in place for 5 minutes then removed. There may be up to 6 treatments (approximately 1 per month).
  Interventions: Drug: Vehicle Patch

INTERVENTIONS:
Drug: VDMN-21 Patch Low Dose — Microneedle patch containing 125 mcg of active drug
  Arms: Treatment Group A (Low Dose)
Drug: VDMN-21 Patch High Dose — Microneedle patch containing 250 mcg of active drug
  Arms: Treatment Group B (High Dose)
Drug: Vehicle Patch — Placebo microneedle patch containing no active drug (i.e., placebo)
  Arms: Treatment Group C (Vehicle)

SUMMARY:
This Phase 2 study has been designed to determine the safety and efficacy of repeated treatment sessions of VDMN-21 patch at two dose strengths as compared to a matched vehicle control patch in subjects with verruca vulgaris

DETAILED DESCRIPTION:
Protocol 250-12951-201 is a planned Phase 2 study entitled "A Multi-Center, Randomized, Double-Blind, Vehicle-Controlled Study of the Safety and Efficacy of VDMN-21 in Subjects with Verruca Vulgaris". Eligible subjects will be randomized into one of the three treatment groups (high dose, low dose, vehicle).

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or non-pregnant female, 9 to 65 years of age.
* Subject has provided written informed consent/assent.
* Females must be post-menopausal, surgically sterile, or use an effective method of birth control. Women of childbearing potential (WOCBP) must have a negative urine pregnancy test (UPT) at Visit 1/Baseline.
* Subject has at least 1 and up to 8 common warts (verruca vulgaris),
* Subject is willing to undergo test article therapy as directed, comply with study instructions (including availability to a smart phone or equivalent device for telehealth visit requirements), and commit to all follow-up visits for the duration of the study.
* Subject is in good general health and free of any disease state or physical condition that might impair evaluation of the identified warts and/or treatment area or exposes the subject to an unacceptable risk by study participation.

Exclusion Criteria:

* Subject is pregnant, lactating, or is planning to become pregnant during the study.
* Subject used or will use oral zinc and/or cimetidine within 30 days prior to enrollment or during the course of the study.
* Subject has received 3 or more prior treatments to the Target Lesion without resolution.
* Subject received any of the following therapies within the specified wash-out period prior to Baseline in the treatment area of the Target Lesion

  1. LASER, light or other energy-based therapy (e.g., intense pulsed light [IPL], PDT; 12 weeks
  2. Immunotherapy (e.g., imiquimod, squaric acid dibutyl ester [SADBE], etc.), retinoids, hydrogen peroxide; 12 weeks
  3. Cryotherapy, biopsy, electrodessication, curettage, antimetabolite therapy (e.g., 5- fluorouracil), cantharidin, or any other treatment that in the opinion of the Investigator may affect the Target Lesion; 6 weeks
  4. Over-the-counter (OTC) wart therapies, paring ± occlusion; 1 week
* Subject has scars, tattoos, or other features that may interfere with the evaluation of the Target Lesion, in the opinion in the investigator.
* Subject has a significant autoimmune condition or is immunocompromised based on their medical condition (e.g., HIV, malignancy, etc.), medication use, or other factors. Routine use of inhaled, intranasal or ophthalmologic corticosteroids during the study is allowed.
* Subject has received systemic immunosuppressive therapy such as steroids, methotrexate, cyclosporine, tacrolimus, chemotherapy, etc. within in 4 weeks prior to Baseline.
* Subject has any active malignancy or are undergoing treatment for any malignancy other than nonmelanoma skin cancer;
* Subject has history of significant ophthalmologic inflammatory disease, including uveitis.
* Subject is currently enrolled in an investigational drug, biologic, or device study.
* Subject has used an investigational drug, investigational biologic, or investigational device treatment within 30 days prior to Visit 1/Baseline.
* Subject has a history of allergy or sensitivity to this antigen extract or similar products.

Ages: 9 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with complete clinical resolution of the Target Lesion at end of treatment period | Baseline up to Day 134
  Complete clinical resolution is defined as the target lesion with area = 0.

OTHER OUTCOMES:
Proportion of subjects with complete clinical resolution of Target Lesion by visit | Days 22, 43, 64, 85, 106, and 134
Proportion of subjects with complete clinical resolution of all the Non-Target Lesion(s) by visit | Days 22, 43, 64, 85, 106, and 134

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Site 07, Fort Smith, Arkansas
  - Site 16, San Diego, California
  - Site 02, Plainfield, Indiana
  - Site 13, Louisville, Kentucky
  - Site 15, Baton Rouge, Louisiana
  - Site 09, New Brighton, Minnesota
  - Site 01, Anderson, South Carolina
  - Site 06, Greenville, South Carolina
  - Site 11, Knoxville, Tennessee
  - Site 03, Arlington, Texas
  - Site 04, Austin, Texas
  - Site 10, College Station, Texas
  - Site 12, Houston, Texas
  - Site 05, Pflugerville, Texas
  - Site 14, Norfolk, Virginia
  - Site 08, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Undecided